CLINICAL TRIAL: NCT03320902
Title: Sudden Death Counselling and Its Impact on Family Members of Sudden Death Victims
Acronym: SUIVIPROCHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: K160905J; 2017-A0098-45 (Other: ID-RCB)
Record Dates: First submitted 2017-10-12; First posted 2017-10-25 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Sudden Death
Keywords: Family members; sudden death; sudden death counseling; depression
MeSH Terms: conditions — Death, Sudden; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sudden death counselling (Active Comparator): The emergency physician of the prehospital EMS who intervenes at the scene will systematically give the family member allocated to the intervention the option to attend a sudden death counselling during the first month after the event.
  Interventions: Behavioral: Sudden death counselling
- Usual practice (No Intervention): The physician will act as usual. The relatives will not systematically benefit from this option.

INTERVENTIONS:
Behavioral: Sudden death counselling — The Sudden Death Counselling with included relatives at 1 month (+/-15 days) after the eventafter the event will be at the Europeen Georges Pompidou hospital in Paris.
  The purpose of this Sudden Death Counselling is to provide to family members of sudden death victims information, support, referral and follow-up services relating to sudden death and their grief, if needed.
  The bereaved people will tell their experience. The Sudden Death Counselling would help them to integrate life's losses by companioning them.
  Cardiologist and psychologists will be present to listen to their pain and try to bring comfort by answering to their questionings.
  Arms: Sudden death counselling

SUMMARY:
Assessment of the psychological benefit of the proposition by prehospital medical team of a sudden death counselling on family members of sudden death victims.

DETAILED DESCRIPTION:
Family members are often shocked and devastated by the death of their loved one, especially when it is sudden and unexpected. On the scene, families often don't really believe it happened because they didn't have time to absorb the fact of their loss. They hear the words and explanation given by the prehospital emergency medical services (EMS) team, but do not comprehend the full impact. Emotions seem frozen. They feel disoriented, restless, stunned and unable to think.

Most often, after cardiac arrest resuscitation attempt, the prehospital EMS team leaves the scene, letting the family without any further medical bond and support. Families are left alone facing this tragedy. After a while, families need medical counseling trying to understand what happens and why but they don't know who to consult. Instead, they remain without medical explanation or guidance with the fear regarding their own future, in particular, regarding the risk of dying from sudden death. This fear may be based on the knowledge of the eventuality of familial diseases increasing the risk of sudden death, or simply on a mechanism of identification with the deceased.

One important factor credited by experts is to encourage first-degree family members to seek sudden death counselling. However, the literature concerning this problem lacks of reliable data.

The aim of this clinical trial is to evaluate the psychological consequences of a sudden death counselling on family member after a relative's sudden death compared to the usual family management.

This study will compare the percentage of depression in a group of family members after a relative's sudden death for whom a sudden death counselling has been proposed by the prehospital medical team versus a group for whom the medical team has not modified its usual strategy.

ELIGIBILITY:
Inclusion Criteria:

A first-degree relative of a:

* patient aged 18-75 years
* with an out-of-hospital sudden death*
* and cardiopulmonary resuscitation attempted Relative aged ≥ 18 years Given consent for the study. Sudden death definition*: An unexpected cardiac arrest without obvious extracardiac cause, leading to a collapse in front of a witness (or in the absence of witnesses, occurring within the hour after the onset of symptoms).

Exclusion Criteria:

Relative under guardianship/curatorship Relative unable to communicate Relative not affiliated to a medical insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 625 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale, sub-section Depression (HADSD) >10 | at 3 months from the sudden death
  Percentage of relatives with moderate to severe symptoms of depression evaluated by the 'Hospital Anxiety and Depression Scale' score, subscale Depression (HADSD) >10
Hospital Anxiety and Depression Scale, sub-section Anxiety (HADSA) >10 | At 3 months from the sudden death
  Percentage of relatives with moderate to severe symptoms of anxiety evaluated by the 'Hospital Anxiety and Depression Scale' score, subscale Anxiety (HADSA) >10

SECONDARY OUTCOMES:
Impact of Event Scale-revised score (IES-R) ≥ 33 | at 3 months from the sudden death
  Percentage of relatives with symptoms of post-traumatic stress disorder evaluated by the 'Impact of Event Scale' score (IES-R) ≥ 33
Medical Outcome Study Short Form Health Survey (SF-12) | At 3 months from the sudden death
  Quality of life questionnaire : the SF-12 is the 12 item abbreviated form of SF-36 survey. It provides information about how participants feel, and how well they have been able to perform their usual activities. SF-12 questions make up 8 scales: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional, Mental Health . Transformed physical component summary score (PCS) and transformed mental component summary score (MCS) are derived using the sum of all 12 items and scored onto a 0-100 scale such that a higher score indicates a better health state and better functioning.
Visits number to the general physician | At 3 months from the sudden death
Drug use | At 3 months from the sudden death
Visits number to the psychologist and/or psychiatrist | At 3 months from the sudden death
Relatives number integrating a grief recovery support group | At 3 months from the sudden death
  Number of participants that have integrated a grief recovery support group
Feeling of the sudden death consultation or not by the relatives | At 3 months from the sudden death
Proportion of identified causes of sudden death | At 3 months from the sudden death
Proportion of familial screening | At 3 months from the sudden death

CONTACTS AND LOCATIONS:
Overall Officials: Patricia JABRE, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants malades, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided